CLINICAL TRIAL: NCT05323448
Title: Efficacy of ARISTA-AH for Restoring Hemostasis Following Posterior Long-segment Spinal Fusion.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinique Bordeaux Nord Aquitaine (Other)
Collaborators: Bard Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-ORT01
Record Dates: First submitted 2022-03-24; First posted 2022-04-12 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hemostatics; Hemostasis; Spinal Deformity; Spinal Fusion
Keywords: ARISTA-TM; Posterior Spinal Fusion; Spinal surgery; Spinal deformity; Hemostasis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARISTA (Experimental): ARISTA-AH will be applied directly within the wound before closure.
  Interventions: Device: ARISTA
- Control group (Experimental): Participant will not receive the ARISTA-AH hemostatic agent.
  Interventions: Device: Control Group

INTERVENTIONS:
Device: Control Group — During the surgical procedure, hemostasis will be achieved using the standard of care (electrocautery, pressure, ligature or any hemostatic agent).
  Arms: Control group
Device: ARISTA — During the surgical procedure, hemostasis will be achieved using the standard of care (electrocautery, pressure, ligature or any hemostatic agent). Before surgical wound closure, the corresponding amount of ARISTA-AH will be applied to completely cover the bleeding site :
  * 5g for 5 to 8 instrumented vertebra
  * 10g fo 9 or more instrumented vertebra
  Arms: ARISTA

SUMMARY:
The aim of this study is to assess the efficacy of the ARISTA AH for restoring hemostasis following a long segment posterior spinal fusion.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written inform consent will be included in the study during their preoperative visit. After eligibility criteria checking and based on their respective surgical indication, participants will be randomized in a single-blinded and stratified manner (participant only) in a 1:1 ratio to ARISTA-AH or no ARISTA-AH. The stratification process will consider the number of instrumented vertebra during each surgery (level 1: 5 to 8 vertebra; level 2: 9 or more instrumented vertebra).

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible to a posterior lumbar or thoraco-lumbar long-segment spinal fusion.
2. Surgery targeting at least 5 adjacent vertebra combined with one of the following procedure:

   1. Intersomatic bone graft;
   2. Pedicle substraction osteotomy;
   3. Any other intervertebral osteotomy (e.g. Smith-Petersen osteotomy);
3. The use of a surgical drain inserted at the operative site is mandatory (suction drain and other drain are eligible);

Exclusion Criteria:

1. Subject under the age of 18 years old;
2. Subject with a known haemostatic disorder;
3. Subject with any infection or any immune system disorder;
4. Subject not eligible to a posterior spinal surgery;
5. Subject with a known allergy or any contraindication to the use of the study device;
6. Currently pregnant or planning pregnancy;
7. Prisoner or a ward of the state;
8. Subject no willing to participate in the study;
9. Subject not affiliated to a social security insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss within the first 24 hours after posterior spinal fusion | 24 hours
  Blood loss calculated in ml per number of instrumented vertebra

SECONDARY OUTCOMES:
Blood loss within the first 6 hours after posterior spinal fusion | 6 hours
  Blood loss calculated in ml per number of instrumented vertebra
Blood loss within the first 48 hours after posterior spinal fusion | 48 hours
  Blood loss calculated in ml per number of instrumented vertebra
Total post-operative blood loss | 3 Days
  Cumulative blood loss observed until surgical drain removal
Estimated Blodd Loss (EBL) | 7 Days
  EBL are calculated by multiplying the perioperative difference of haemoglobin EHb (formula used: EHb = (Hb preop - Hb post-op)/Hb preop) by the patient's estimated blood volume (EBV = weight x F; F = 75 for adult males; F = 70 for adolescent males; F = 60 for females).
  EBL = EHb x EBV
Hidden Blood Loss (HBL) | 7 Days
  HBL is the difference of the estimated blood loss (EBL) with the amount of perioperative blood loss and the amount of transfusions:
  HBL = EBL - intraoperative blood loss + transfusion
Drain removal | 7 Days
  Delay between the date of initial surgery and the date of surgical drain removal
Detection of any early post-operative haematoma | 7 Days
  Every participant will have an early postoperative MRI (before hospital discharge) to detect the presence of any haematoma.
  The presence (yes/no), the size (cm2) and the gravity (symptomatic, asymptomatic) of the observed haematoma will be compared between the 2 groups
Improvement of back and leg pains at 3 months compared to preoperative scores | 3 months
  Back and leg pain intensity self-report will be assessed before and after initial procedure for each patient (at 3 months) using a 0 to 10 visual analog scale (0: no pain ; 10: most imaginable pain).
Assessment of the Oswestry Disability Index | 3 months
  Change from baseline in self reported Oswestry Disability Index (ODI) score at 3 months.
Change in Patient's quality of life | 3 months
  Change from baseline in self reported 12-Item Short Form Survey (SF-12) score at 3 months.
Length of stay | 7 Days
  Length of stay is the delay between the date of admission and the date of discharge for each patient.
Detection of any haemostasis disorder | 3 Months
  Proportion of subjects with any of the following complications related to haemostasis condition: delay or healing disorders, post-operative wound infection, neurological disorders, surgical disorders or any other complication directly related to haemostasis dysfunction or the use of ARISTA-AH product.
Incidence of any serious adverse events | 3 Months
  Record of any intra and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jean Charles LE HUEC, M.D., PhD, Principal Investigator — VERTEBRA Institute, Polyclinique Bordeaux Nord Aquitaine
Locations (1):
- Polyclinique Bordeaux Nord Aquitaine, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No